CLINICAL TRIAL: NCT05805865
Title: Efficacy of Eco-Friendly Toothpaste Tablets Versus Conventional Toothpaste Using PI and GI Index
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5220342
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Gingival Inflammation
Keywords: Gingival Index; Plaque Index; Dentifrice; Toothpaste Tablets; Consumer Satisfaction
MeSH Terms: conditions — Gingivitis; Consumer Behavior | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator blinded to group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Toothpaste Tablet (Experimental): Subjects are instructed to use one toothpaste tablet for brushing. Brushing is recommended twice daily for two minutes.
  Interventions: Drug: Toothpaste Tablet
- Conventional Toothpaste (Active Comparator): Subjects are instructed to use the toothpaste for brushing. Brushing is recommended twice daily for two minutes.
  Interventions: Drug: Conventional Toothpaste

INTERVENTIONS:
Drug: Toothpaste Tablet — Colgate Anywhere Toothpaste Tablets
  Arms: Toothpaste Tablet
Drug: Conventional Toothpaste — Colgate Cavity Protection
  Arms: Conventional Toothpaste

SUMMARY:
Objectives: To assess the change in gingival index (GI) and plaque index (PI) when comparing the use of toothpaste tablets to conventional toothpaste.

Methods: 40 participants were randomized into two groups: Colgate's toothpaste tablets (T) and Colgate's Cavity Protection toothpaste (C). Both groups utilized their assigned dentifrice for 2 weeks. A pre and post-assessment measured the GI and PI index. A questionnaire on the use of the product was distributed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 18 years or older;
2. Subjects who will comply with study protocol;
3. Subjects who can read and understand the consent form;
4. Subjects available during the study period;
5. Subjects have more than 20 teeth.

Exclusion Criteria:

1. Subjects who are pregnant and/or nursing;
2. Subjects under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Kwon, DDS, MS, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toothpaste Tablet | Conventional Toothpaste
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toothpaste Tablet | Conventional Toothpaste | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.95 (4.20) | 25.35 (4.15) | 25.15 (4.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index Score at Baseline
Description: Plaque was scored according to the Turesky modification of the Quigley-Hein Plaque Index. Each tooth was divided into six surfaces, three facial and three lingual, as follows: 1) mesio-facial; 2) mid-facial; 3) disto-facial; 4) mesio-lingual; 5) mid-lingual; and 6) disto-lingual. Teeth included in the scoring were: #3, 7, 12, 19, 23, 28. Plaque was disclosed and scored on each tooth surface according to the following criteria:
  0: No plaque.
  1. Separate flecks of plaque at the cervical margin.
  2. A thin, continuous band of plaque (up to 1 mm) at the cer- vical margin.
  3. A band of plaque wider than 1 mm but covering less than 1/3 of the side of the crown of the tooth.
  4. Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth.
  5. Plaque covering 2/3 or more of the side of the crown of the tooth.
  Subject-wise scores were determined by averaging the values obtained over all scorable surfaces in the mouth.
Time Frame: Change between baseline at visit 1 and visit 2, two weeks post baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Toothpaste Tablet | Conventional Toothpaste
Number analyzed (Participants) | 20 | 20
Score on a scale | 2.80 (0.58) | 2.78 (0.46)

2. Primary Outcome: Gingival Index Score at Baseline
Description: Gingivitis was scored according to the Löe-Silness Gingival Index. Each tooth was divided into six surfaces, three facial and three lingual, as follows: 1) mesio-facial; 2) mid-facial; 3) disto-facial; 4) mesio-lingual; 5) mid-lingual; and 6) disto-lingual. Teeth included in the scoring were: #3, 7, 12, 19, 23, 28. The gingiva adjacent to each tooth surface was scored as follows:
  0 = Absence of inflammation.
  1. = Mild inflammation-slight change in color and little change in texture.
  2. = Moderate inflammation-moderate glazing, redness, edema, and hypertrophy.
  3. = Severe inflammation-marked redness and hypertrophy. Tendency for spontaneous bleeding.
  Subject-wise scores were determined by averaging the values obtained over all scorable surfaces in the mouth.
Time Frame: Change between baseline at visit 1 and visit 2, two weeks post baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Toothpaste Tablet | Conventional Toothpaste
Number analyzed (Participants) | 20 | 20
Score on a scale | 1.35 (0.26) | 1.37 (0.24)

3. Secondary Outcome: Subject Perception of Product Use
Description: This is a composite measurement based on questionnaire response. Subjects will answer 7 questions related to cleanliness, flavor, ease of use, eco-friendliness, willingness to switch, satisfaction, texture. This is measured on a Likert Scale from 1-4. 1 represents strongly agree with overall product satisfaction. 4 represents strongly disagree with overall product satisfaction.
Time Frame: Visit 2 two weeks post study enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste Tablet | Conventional Toothpaste
Number analyzed (Participants) | 20 | 20
units on a scale | 2.0 (0.4) | 1.7 (0.4)

ADVERSE EVENTS:
Time Frame: Two weeks post-baseline
Arm/Group | Toothpaste Tablet | Conventional Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT05805865/Prot_SAP_000.pdf